CLINICAL TRIAL: NCT06408480
Title: Neonatologist-performed Lung Ultrasound During Immediate Transition After Birth to Predict the Need for Respiratory Support Persisting More Than 1 Hour - a Pilot Study
Brief Title: Neonatologist-performed Lung Ultrasound in the Delivery Room
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 36-150 ex 23/24
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Disease
Keywords: neonatologist-performed lung ultrasound; postnatal transition; neonates
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- need of respiratory support > 60 min after birth: Group comprises neonates in need of further respiratory support more than 60 minutes after birth.
  Interventions: Diagnostic Test: Neonatologist-performed lung ultrasound
- need of respiratory support < 60 min after birth: Group comprises neonates that show any signs of respiratory distress in the first 60 minutes, but do not need respiratory support more than 60 minutes after birth.
  Interventions: Diagnostic Test: Neonatologist-performed lung ultrasound

INTERVENTIONS:
Diagnostic Test: Neonatologist-performed lung ultrasound — lung ultrasound conducted in min 5, 15, 30, 60 min after birth in late preterm and term infants

SUMMARY:
The objective of this study is to evaluate the role of the neonatologist-performed lung ultrasound (NPLUS) during immediate transition after birth of late preterm and full-term neonates using the lung ultrasound score to predict the need of respiratory support persisting more than 1 hour after birth.

DETAILED DESCRIPTION:
Lung ultrasound is an emerging clinical tool to assess the lung in a dynamic way. Recently, the focus has been on establishing lung ultrasound in the neonatal intensive care unit (NICU) as a point-of care application.

Neonates born by a Caesarean section are particularly prone to have an altered adaption to extrauterine life. Especially in the first hours after birth, respiratory distress syndromes (RDS) may occur due to delayed lung fluid clearance after birth.

While acute RDS in the first hours after birth may be a self-limiting disorder and therefore a benign condition, it remains difficult to identify neonates in need for further respiratory support at the NICU. Admission to the NICU not only causes parental stress but also contributes to additional healthcare costs.

There is emerging evidence that NPLUS is a reliable tool to differentiate between the causes leading to RDS in neonates. Using a neonatologist performed lung ultrasound score for the early identification of neonates in need of respiratory support persisting more than 1 hour would be therefore highly advantageous.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm neonates (born between 34 0/7 and 36 6/7 weeks of gestation) and full-term neonates (born later than 36 6/7 weeks of gestation) delivered by Caesarean section
* Presence of any sign of respiratory distress (defined as tachypnoea/ dyspnoea, grunting, flaring of the nostrils or chest retractions)
* Written informed consent obtained from the parents prior to birth.

Exclusion Criteria:

* Presence of cardiopulmonary malformations
* Patients with pneumothorax diagnosed by neonatologist-performed lung ultrasound

Max Age: 60 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Late preterm neonates (born between 34 0/7 and 36 6/7 weeks of gestation), and full-term neonates (born later than 36 6/7 weeks of gestation) delivered by Caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the change in lung ultrasound score according to Rodriguez-Fanjul et al. 2020 | 60 minutes for all scans, 2-4 min per scan.
  Score determined by neonatologist-performed lung ultrasound conducted at 5, 15, 30 and 60 minutes after birth. The lung ultrasound score will be calculated by performing bilateral longitudinal scans of the chest on the midclavicular, anterior, and posterior axillary line.
  For every scan a score is given ranging from 0 (for normal lung aeration) up to 3 (describing extended consolidations in the lung).
The need for respiratory support persisting more than 1 hour after birth | 60 minutes
  binary - yes/ no
Admission to the Neonatal Intensive Care Unit | 60 minutes
  binary - yes/ no

SECONDARY OUTCOMES:
Length of respiratory support | 60 minutes
  in minutes
Mode of respiratory support | 60 minutes
  non-invasive versus invasive ventilation
Routinely obtained capillary blood gas analysis of the newborn | 60 minutes
  pCO2, pO2, pH, BE, HCO3, lactate, glucose
Routinely obtained monitoring parameters- SpO2 | 60 minutes
  arterial oxygen saturation (SpO2)
Routinely obtained monitoring parameters- heart rate | 60 minutes
  heart rate in beats per minute (either by pulse oximetry or electrocardiography)
Routinely obtained monitoring parameters- cerebral oxygen saturation | 60 minutes
  cerebral oxygen saturation (assessed by near-infrared spectroscopy)
SpO2/FiO2 | 60 minutes
  fraction of inspired oxygen ratio to O2 supply
pH of the umbilical artery | 15 minutes
  in numbers
APGAR score | 10 minutes
  Score ranges from 0 to 10, higher score indicates a better outcome
Number of Participants with Presence of pregnancy risk factors | 10 minutes
  including intra-amniotic infection, and premature rupture of the membranes
Number of Participants with Prenatal corticosteroids | 10 minutes
  binary - yes/ no

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwaberger, MD PhD, Principal Investigator — Division of Neonatology, Medical University of Graz, Austria
Locations (1):
- Division Neonatology, Dp. Pediatrics, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT06408480/Prot_SAP_000.pdf